CLINICAL TRIAL: NCT02686008
Title: A Pilot Pharmacodynamic Study to Assess the Anti-proliferative Activity a of the Poly ADP Ribose Polymerase (PARP) Inhibitor Olaparib in Patients With Human Papilloma Virus (HPV) Positive and Human Papilloma Virus (HPV) Negative Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Pharmacodynamic Study to Assess the Anti-proliferative Activity of the PARP Inhibitor Olaparib in Patients With HPV Positive and HPV Negative HNSCC
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was stopped due to lack of funding.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1409014536
Record Dates: First submitted 2015-09-24; First posted 2016-02-19 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HPV negative tumors (Experimental): 10 patients with HPV negative tumors: Non-oropharyngeal tumors or p16 negative and HPV negative oropharyngeal tumors
  Interventions: Drug: Olaparib
- HPV positive tumors (Experimental): 10 patients with HPV positive tumors: p16 positive and HPV positive tumors
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Patients will receive olaparib administered at 300 mg bid x 14 days orally
  Other Names: Lynparza

SUMMARY:
This is an open label pilot study evaluating the pharmacodynamics and safety of single agent olaparib administered at 300mg bid (twice a day) for 14 days orally in patients with human papillomavirus (HPV) -positive and human papillomavirus (HPV)-negative head and neck squamous cell carcinoma (HNSCC)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HNSCC with surgically resectable disease
* No prior chemotherapy or radiation therapy as treatment for the observed HNSCC
* Patients must provide written informed consent
* Age >=18 years of age
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of <2
* Normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:
* Hemoglobin >= 10 g/dL and no blood transfusions in the 28 days prior to entry/randomization
* Absolute neutrophil count >=1.5 x 10^9/L
* No features suggesting of MDS/AML on peripheral blood smear
* White blood cells > 3 x 10^9/L
* Platelet count >= 100 x 10^9/L
* Total bilirubin <= 1.5 x institutional upper limit of normal (ULN)
* AST (SGOT)/ALT (SGPT) < 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be < 5x ULN
* Serum creatinine <= 1.5 x institutional ULN OR creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of the study participation and must have negative serum or urine pregnancy test within 1 week prior to beginning treatment on this trial
* Must be abler to understand and sign a written informed consent document

Exclusion Criteria:

* Patients with known brain metastases. Patients may have received WBRT within 14 days or focal radiation within 1 week of cycle 1, day 1. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 28 days prior to treatment
* Women must not be pregnant or breastfeeding
* Patients with known hypersensitivity to olaparib or any of the excipients of the product
* Patients receiving any other investigational agents within 4 weeks of starting the study
* Involvement in the planning and/or conduct of the study
* Any previous treatment with a PARP inhibitor, including olaparib
* Concomitant use of known CYP3A4 inhibitors such as ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin, and nelfinavir
* Persistent toxicities (>=CTCAE grade 2)
* Resting ECG with QTC >470msec on 2 or more time points within a 24 hour period or family history of long QT syndrome
* Blood transfusions within 1 month prior to study start
* Patients with myelodysplastic syndrome/acute myeloid leukemia
* Major surgery within 14 days of starting study treatment and patients must have recovered from any effects of any major surgery
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection.
* Unable to swallow oral medication
* Immunocompromised patients, e.g., patients who are known to be serologically positive for HIV and are receiving antiviral therapy
* Known active hepatic disease
* Uncontrolled seizures
* Previous cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for 5 years
* Currently on warfarin(subcutaneous heparin is permitted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Change in Level of IHC-Ki-67 expression | Baseline and 14 days
  Tissue biopsy sections will be analyzed for proliferation (IHC-Ki-67) Ki-67 is a nuclear non-histone protein that is present at low levels in quiescent cells but is increased in proliferating cells. Thus, Ki-67 reactivity, defined as percent tumor cells staining positive as measured by immunohistochemical (IHC) staining, is a specific nuclear marker for cell proliferation.

SECONDARY OUTCOMES:
Change in Tissue apoptosis | Baseline and 14 days
  Tissue biopsy sections will be analyzed for apoptosis. For example using the IHC-cleaved caspase-3 assay.
Change in DNA repair pathways | Baseline and 14 days
  Tissue biopsy sections will be analyzed to determine effect on DNA repair pathways (PARP activity). Specifically Poly(ADP-ribose) immunohistochemical staining of tissue biopsies will be performed and PAR intensity scored as 0 (no signal), 1 (weak), 2 (strong intensity in >50% of tumor cells).

CONTACTS AND LOCATIONS:
Overall Officials: Anne Chiang, MD, PhD, Principal Investigator — Yale University